CLINICAL TRIAL: NCT00435474
Title: Malignant Wounds: A Randomized Clinical Trial Investigating a Complementary Multidimensional Intervention
Brief Title: Malignant Wounds, Wound Treatment, Psycho-Social Support and Relaxation Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: kf 0102006-5491
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Last update posted 2009-06-09 (Estimated); Status verified 2009-06

CONDITIONS: Cancer; Malignant Wounds
Keywords: Cancer; Malignant wounds; Quality of life; Body-Image; Cancer patients
MeSH Terms: conditions — Neoplasms | interventions — Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Silver product
  Interventions: Procedure: Wound treatment; Other: psycho-social support; Other: relaxation therapy
- 2 (Experimental): Honey product
  Interventions: Procedure: wound treatment; Other: psycho-social support; Other: relaxation therapy

INTERVENTIONS:
Procedure: Wound treatment — wound treatment (silver product, alginate and foam dressing)
  Arms: 1
Procedure: wound treatment — wound treatment (honey product, alginate and foam dressing)
  Arms: 2
Other: psycho-social support — psycho-social support (based on the structure in cognitive therapy)
Other: relaxation therapy — relaxation therapy

SUMMARY:
The purpose of this study is to investigate whether treatment for cancer patients with malignant wounds can improve (wound healing/wound size, odor, infection, seepage, pain) through comparing the effects of two multidimensional interventions including wound treatment, psycho-social support and relaxation therapy.

DETAILED DESCRIPTION:
Objective: To investigate whether treatment for cancer patients with malignant wounds can improve (wound healing/wound size, odor, infection, seepage, pain) through comparing the effects of two multidimensional interventions:

1. wound treatment (silver product, alginate and foam dressing >< honey product, alginate and foam dressing) in combination with,
2. psycho-social support (based on the structure in cognitive therapy) and
3. relaxation therapy.

Furthermore to investigate coping strategies, body image, stigma and quality of life in cancer patients with malignant wounds.

Design: A hypothesis testing prospective randomized clinical intervention study (n=70) and an explorative qualitative interview study

Method: Digital photographing, measurement of wound size with Quantify-Image-One, wound morphology registration (the extent of malodour, infection, seepage, bleeding, pain, the healing process), grafting, VAS-score, quality of life questionnaire (EORTC-QLQ-C30, DLQI), Hospital Anxiety and Depression Scale (HAD), Mental Adjustment to Cancer (MAC), interview.

Patients will fill out a diary focusing on wound related problems.

Perspectives: The results will determine whether the honey treatment is an improvement, and whether the silver treatment has statistical and clinical significance.

The qualitative study will contribute new knowledge about conditions of life for cancer patients with cancer wounds, their feelings and impositions.

In spite of proving positive effect, the project will contribute with new required knowledge on treatment and support for cancer patients suffering from malignant wounds.

ELIGIBILITY:
Inclusion Criteria:

* Cancer with evidence of disease.
* Cancer wound >2 cm.
* Receiving antineoplasm treatment.
* > 18 years.
* Receiving antineoplasm treatment in out-patient clinic.
* Read, speak and write Danish.

Exclusion Criteria:

* No radiation therapy the last 6 month (on the wound).
* Life expectancy > 3 month.
* Not psychotic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Wound size | after four weeks intervention period

SECONDARY OUTCOMES:
Wound odor. Wound infection. Wound exudate. Wound pain. Anxiety and depression. Body-Image.Sexuality.Quality of life. | after the four week intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Lis Adamsen, Professor, Study Chair — Copenhagen University. Faculty of health Sciences, Denmark
Locations (1):
- Rigshospitalet, University hospital of Copenhagen. Oncology department, Copenhagen, Denmark